CLINICAL TRIAL: NCT05950217
Title: The Effect of Preoperative Education on Kinesiophobia in Patients Undergoing Total Knee Replacement Surgery: A Randomized Controlled Study
Brief Title: Kinesiophobia in Patients Undergoing Total Knee Replacement Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Bahar CANDAS ALTINBAS, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nurse_Kinesiophobia02
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Kinesiophobia
Keywords: Kinesiophobia; Knee replacement; Nursing education; Preoperative care
MeSH Terms: conditions — Kinesiophobia | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group patients will be educated by the nurse in the preoperative period with the support of visual education material
  Interventions: Other: Education
- Control Group (No Intervention): The control group will take rutin patient care.

INTERVENTIONS:
Other: Education — Nurse-led patient education
  Arms: Experimental Group

SUMMARY:
Providing information to the patient before surgery has important effects on the patient's self-care skills regarding the treatment and care process, reducing stress and reducing fears in the postoperative period. The primary aim of this study was to examine the effect of preoperative education on kinesiophobia in patients undergoing total knee replacement surgery. In addition, preoperative anxiety levels, time of first postoperative mobilization, number of steps in the first 24 hours after mobilization and pain levels of the patients will be evaluated as secondary outcomes.

DETAILED DESCRIPTION:
Kinesiophobia is known as the minimization of activities or avoidance of movement due to the fear that the pain caused by movement will negatively affect the person's life and the problem will occur again. It was first defined by Miller, Kopri and Todd in 1990 at the American Pain Society meeting as excessive and unreasonable anxiety against physical movement and pain in the person, which occurs due to the person feeling vulnerable as a result of a painful injury or re-injury. Kinesiophobia is one of the factors that contribute to the chronicization of pain in individuals after surgery; it can lead to negative patient behaviors on the disease in the surgical process. In addition, kinesiophobia can lead to movement limitation and movement limitation can lead to pain. Since this vicious cycle may result in more pain and disability, the importance of the issue is increasing. It has also been shown that patients with high levels of kinesiophobia experience more pain and have a lower quality of life. This research project aims to provide an original approach in a field where studies on preventing or minimizing the effects of kinesiophobia on the surgical process and postoperative recovery process are limited. It is expected that nurses' interventions for kinesiophobia during the operation process will have positive effects on treatment and care. In this study, visual material-supported patient education will be provided to reduce the level of kinesiophobia associated with total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Planned surgery
* Speaking and understanding Turkish
* Being admitted to the hospital at least one day before the surgery

Exclusion Criteria:

* Visual, hearing and speech disabilities,
* Being mentally disabled,
* Having a psychiatric disorder or being in the process of treatment
* Having had knee replacement surgery before

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-05-29 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | 2 days
  Self reported kinesiophobia intensity after surgical process that includes one day after surgery. TAMPA Kinesiophobia Scale (TSK) will be used to evaluate the kinesiophobia. The TSK consists of 17 items that are rated on a 4-point Likert scale, ranging from "Strongly Disagree" to "Strongly Agree." It is scored by assigning a numerical value to each response. Individual item scores range from 1-4, with the negatively worded items (4,8,12,16) having a reverse scoring (4-1). The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.

SECONDARY OUTCOMES:
Anxiety level | 2 days
  Self reported anxiety intensity before surgical process that includes on the day of surgery. State-Trait Anxiety Inventory will be used to evaluate the anxiety. The higher the score is the more anxiety.
Pain level | 1 day
  It means that what is the severity of the pain that the patients had in 24 hours after surgery. It evaluated with Visual Analog Scale. The most common style used in pain measurement uses a horizontal line measuring exactly 10 cm. The patient is asked to make a mark on this line (from 0 to 10), then the line is measured and recorded in millimeters or centimeters. The higher the score is the more severe the pain. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
First postoperative mobilization time | 1 day
  How many hours after surgery did the patients walk for the first time? This metric will be recorded as day using a questionnaire. The minimum, maximum, median, 25th, and 75th quartiles were calculated for each group and compared. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
Number of steps in the first 24 hours after mobilization | 1 day
  How many steps did the patients take in 24 hours after surgery? This parameter will be evaluated with a pedometer bracelet to be worn on the arm of the patients. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Candas Altinbas, PhD, Principal Investigator — Karadeniz Technical University
Locations (2):
- Turkey (Türkiye) (2):
  - Bahar Candas Altinbas, Trabzon
  - Nurdan Reis, Trabzon

IPD SHARING:
Plan to Share IPD: No